CLINICAL TRIAL: NCT06312969
Title: Cognitive Training Through Technological Gaming To Ameliorate Cognitive Effects Related To Childhood Cancer Treatment (WINNERS)
Brief Title: Technological Gaming in Cancer Survivors (WINNERS)
Acronym: WINNERS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Antonio Pérez Martínez (Other)
Collaborators: Hospital Ruber Internacional (Other); Universidad Rey Juan Carlos (Other)
Responsible Party: Sponsor-Investigator, Antonio Pérez Martínez, Head of the Hemato-Oncology department, Instituto de Investigación Hospital Universitario La Paz
Organization: Instituto de Investigación Hospital Universitario La Paz (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022.301
Record Dates: First submitted 2023-06-09; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Survivors of Childhood Cancer
Keywords: Cancer Survivors; Survivors of Childhood Cancer; Chemotherapy-related Cognitive Impairment; Functional Magnetic Resonance Imaging (fMRI); Video Games; Exergaming
MeSH Terms: conditions — Chemotherapy-Related Cognitive Impairment

STUDY DESIGN:
Intervention Model Description: Randomized versus control group clinical trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group with video game-based training (Experimental): Cognitive training through 3 types of video games:
  * "Serious games" or "brain-training games".
  * Exer-gaming
  * Skill-training games Method of administration
  The patient will receive the treatment for a period of 12 weeks, in which they will commit to use the video games of the intervention with the following pattern:
  * "Brain-training game": sessions of 7-12 minutes with a frequency of 4 days a week.
  * "Exer-gaming": sessions of 15-20 minutes 2 days a week.
  * "Skill-training games": sessions of 15-20 minutes 2 days a week.
  Interventions: Behavioral: Video game based training
- Waiting group (no training) (No Intervention): Patients in waiting group will not receive treatment whilst the 3 month period.

INTERVENTIONS:
Behavioral: Video game based training — Type of intervention: Cognitive training through 3 types of video games:
  * "Serious games" or "brain-training games".
  * Exer-gaming
  * Skill-training games
  Method of administration: The patient will receive the treatment for a period of 12 weeks, in which they will commit to use the video games of the intervention with the following pattern:
  * "Brain-training game": sessions of 7-12 minutes with a frequency of 4 days a week.
  * "Exer-gaming": sessions of 15-20 minutes 2 days a week.
  * "Skill-training games": sessions of 15-20 minutes 2 days a week.
  Arms: Intervention group with video game-based training

SUMMARY:
HYPOTHESIS

1. Neurocognitive deficits in cancer survivors are underestimated. They represent a very limiting long-term side effect in this group of patients.
2. An individualized, planned and limited intervention using technological gaming can improve neurocognitive function in these pediatric patients by taking advantage of the plasticity of the central nervous system (CNS) in the pediatric age.
3. Changes can be demonstrated not only at the cognitive level, but also at the structural and functional level using neuroimaging techniques after our intervention.
4. In addition to the aforementioned benefits, this therapeutic tool can improve some clinical-analytical markers used in the follow-up of cancer survivors, such as immunological markers like lymphocyte populations and inflammatory cytokines.
5. The neurocognitive effects of this therapy are not only produced at the time of the intervention, but remain until months after the intervention.
6. The positive impact of the treatment is not only observed in the patients, but also in the psychological and emotional state of the family members.

VARIABLES

1. Clinically relevant improvement with moderate or large effect size in the following parameters as measured by neuropsychological tests.
2. Statistically significant changes in neuroimaging tests.
3. Statistically significant changes in immune and inflammatory biomarkers before and after treatment.

STUDY DESIGN In this clinical trial, randomized versus control group, unblinded, the aim is to demonstrate the neuropsychological, structural and functional benefit of an intervention using video games in child cancer survivors.

POPULATION OF THE STUDY The target population participating in the study will include patients of either sex aged 8-17 years who completed cancer treatment 1-5 years ago. They must have received treatment with neurotoxic potential: intrathecal/intraventricular chemotherapy, high-dose chemotherapy with crossing of the blood-brain barrier, CNS radiotherapy or hematopoietic stem cell transplantation (HSCT).

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE Several authors have described specific cognitive damage following cancer treatments (often chemotherapy and radiotherapy), which has been termed "chemo-brain". This condition produces alterations in different neurocognitive fields such as memory, learning, concentration, reasoning, executive functions, attention and visuospatial skills.

In this research project the investigator team propose an intervention aimed at one of the most limiting adverse effects of cancer and its treatment such as neurocognitive deficits through technological game platforms and brain training used in a directed, controlled and supervised manner.

HYPOTHESIS

1. Neurocognitive deficits in cancer survivors are underestimated. They represent a very limiting long-term side effect in this group of patients.
2. An individualized, planned and limited intervention using technological gaming can improve neurocognitive function in these pediatric patients by taking advantage of the plasticity of the central nervous system (CNS) in the pediatric age.
3. Changes can be demonstrated not only at the cognitive level, but also at the structural and functional level using neuroimaging techniques after our intervention.
4. In addition to the aforementioned benefits, this therapeutic tool can improve some clinical-analytical markers used in the follow-up of cancer survivors, such as immunological markers like lymphocyte populations and inflammatory cytokines.
5. The neurocognitive effects of this therapy are not only produced at the time of the intervention, but remain until months after the intervention.
6. The positive impact of the treatment is not only observed in the patients, but also in the psychological and emotional state of the family members.

VARIABLES

1. Clinically relevant improvement with moderate or large effect size in the following parameters as measured by neuropsychological tests: TAVECI/TAVEC, CATA, TONI-4 (form A), Digits, SDMT, ROCF, TFV, Stroop, Vocabulary
2. Statistically significant changes in neuroimaging tests. The following variables will be measured:

   1. Structural imaging: volume measurement and Voxel Based Morphometry
   2. Diffusion Imaging: diffusion maps and structural connectivity
   3. Functional imaging: resting state and task based fMRI
3. Statistically significant changes in immune and inflammatory biomarkers before and after treatment:

   1. Study of lymphocyte populations by parametric flow cytometry: T lymphocytes, B lymphocytes, natural killer (NK) lymphocytes, NK T lymphocytes
   2. Study of inflammatory cytokines by LUMINEX: IL-2, IL-4, IL-6, TNF alpha, IFN gamma, IL-10, IL-17TH, IL-1R antagonist

STUDY DESIGN

In this clinical trial, randomized versus control group, unblinded, the aim is to demonstrate the neuropsychological, structural and functional benefit of an intervention using video games in child cancer survivors, patients will follow the following phases:

* Informed consent
* Recruitment, inclusion and exclusion criteria.
* Initial T0 assessment
* Randomization
* Treatment phase for the intervention group. Waiting phase for control group
* Early post-treatment evaluation T+3
* Late post-treatment evaluation T+6

POPULATION OF THE STUDY The target population participating in the study will include patients of either sex aged 8-17 years who completed cancer treatment 1-5 years ago. They must have received treatment with neurotoxic potential: intrathecal/intraventricular chemotherapy, high-dose chemotherapy with crossing of the blood-brain barrier, CNS radiotherapy or hematopoietic stem cell transplantation (HSCT).

TREATMENT OF THE STUDY Type of intervention

Cognitive training through 3 types of video games:

* "Serious games" or "brain-training games".
* Exer-gaming
* Skill-training games Method of administration

The patient will receive the treatment for a period of 12 weeks, in which they will commit to use the video games of the intervention with the following pattern:

* "Brain-training game": sessions of 7-12 minutes with a frequency of 4 days a week.
* "Exer-gaming": sessions of 15-20 minutes 2 days a week.
* "Skill-training games": sessions of 15-20 minutes 2 days a week.

SAMPLE SIZE It is planned to recruit 56 patients (28 patients for each group, of which 14 will be from the 8-12 years age group and 14 will be from the 13-17 years age group). Recruitment will be for 12 months, with a follow-up period for each patient of 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 8 and 17 years of age at the time of recruitment.
* Have completed treatment between 1 and 6 years prior to recruitment.
* Have had one of the following diagnoses:

  * Patients with CNS disease (posterior fossa tumors and supratentorial gliomas smaller than 1 cm affecting associative areas).
  * Patients with hematologic malignancies (leukemia or lymphoma).
  * Patients with solid tumors.
  * Patients with non-malignant hematological diseases and indication for allogeneic hematopoietic progenitor transplantation.
* Having received at least one of the following treatments:

  * Central nervous system surgery.
  * Central nervous system radiotherapy.
  * Intrathecal/intraventricular chemotherapy.
  * Neurotoxic systemic chemotherapy.
  * Hematopoietic stem cell transplantation.
* Informed consent signed by parent/guardian.

Exclusion Criteria:

* Active oncologic disease or relapse of active oncologic disease.
* Prior neurological or psychiatric pathology that may preclude trial or treatment evaluations:

  * Psychological or neurocognitive illness or sequelae that preclude neuropsychological assessment or are expected to significantly artifact MRI results (examples: significant decrease in visual acuity, CNS surgical scar that artifacts imaging results, severe cognitive delay that precludes testing, etc.).
  * Psychological or neurocognitive illnesses or sequelae that prevent or contraindicate the use of video games (epilepsy that prevents the use of screens, significant decrease in visual acuity, etc.).
  * Mild or self-limiting neurological or psychiatric pathology that does not interfere with trial diagnosis and treatment (headache, epilepsy in remission with effective treatment, mild cognitive delay, etc.) will be allowed.
* Current or recent (less than 1 year) use of other cognitive stimulation or brain training that may interfere with study results.
* Refusal to abstain from the use of the study treatment games in case of being assigned to group B (control group).
* Medical treatment that may significantly interfere with neuropsychological, imaging or biomarker assessments.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 56 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
SDMT Test | Baseline
  To evaluate the benefits of treatment at the neurocognitive level by means of neuropsychological tests.
Change in SDMT Test | At 3 months after recruitment
  To evaluate the benefits of treatment at the neurocognitive level by means of neuropsychological tests.
Change in SDMT Test | At 6 months after recruitment
  To evaluate the benefits of treatment at the neurocognitive level by means of neuropsychological tests.
"DIGITOS" Test | Baseline
  To evaluate the benefits of treatment at the neurocognitive level (processing speed)
Change in "DIGITOS" Test | At 3 months after recruitment
  To evaluate the benefits of treatment at the neurocognitive level (processing speed)
Change in "DIGITOS" Test | At 6 months after recruitment
  To evaluate the benefits of treatment at the neurocognitive level (processing speed)
"TONI-4" test | Baseline
  To evaluate the benefits of treatment at the neurocognitive level (non-verbal intelligence)
Change in "TONI-4" test | At 3 months after recruitment
  To evaluate the benefits of treatment at the neurocognitive level (non-verbal intelligence)
Change in "TONI-4" test | At 6 months after recruitment
  To evaluate the benefits of treatment at the neurocognitive level (non-verbal intelligence)
"ROCF" test | Baseline
  To evaluate the benefits of treatment at the neurocognitive level (visuo-constructional ability and non-verbal memory)
Change in "ROCF" test | At 3 months after recruitment
  To evaluate the benefits of treatment at the neurocognitive level (visuo-constructional ability and non-verbal memory)
Change in "ROCF" test | At 6 months after recruitment
  To evaluate the benefits of treatment at the neurocognitive level (visuo-constructional ability and non-verbal memory)
"TFV" test | Baseline
  To evaluate the benefits of treatment at the neurocognitive level (verbal fluency)
Change in "TFV" test | At 3 months after recruitment
  To evaluate the benefits of treatment at the neurocognitive level (verbal fluency)
Change in "TFV" test | At 6 months after recruitment
  To evaluate the benefits of treatment at the neurocognitive level (verbal fluency)
"STROOP" test | Baseline
  To evaluate the benefits of treatment at the neurocognitive level (selective attention and inhibitory control)
Change in "STROOP" test | At 3 months after recruitment
  To evaluate the benefits of treatment at the neurocognitive level (selective attention and inhibitory control)
Change in "STROOP" test | At 6 months after recruitment
  To evaluate the benefits of treatment at the neurocognitive level (selective attention and inhibitory control)
"TAVECI" test | Baseline
  To evaluate the benefits of treatment at the neurocognitive level (verbal learning)
Change in "TAVECI" test | At 3 months after recruitment
  To evaluate the benefits of treatment at the neurocognitive level (verbal learning)
Change in "TAVECI" test | At 6 months after recruitment
  To evaluate the benefits of treatment at the neurocognitive level (verbal learning)
"CPT3" | Baseline
  To evaluate the benefits of treatment at the neurocognitive level (performance in attention tasks)
Change in "CPT3" | At 3 months after recruitment
  To evaluate the benefits of treatment at the neurocognitive level (performance in attention tasks)
Change in "CPT3" | At 6 months after recruitment
  To evaluate the benefits of treatment at the neurocognitive level (performance in attention tasks)
"BRIEF" survey | Baseline
  To evaluate the benefits of treatment at the neurocognitive level (assessment of executive functions by parents)
Change in "BRIEF" survey | At 3 months after recruitment
  To evaluate the benefits of treatment at the neurocognitive level (assessment of executive functions by parents)
Change in "BRIEF" survey | At 6 months after recruitment
  To evaluate the benefits of treatment at the neurocognitive level (assessment of executive functions by parents)
"BASC" survey | Baseline
  To evaluate the benefits of treatment at the neurocognitive level (Behavior Assesment)
Change in "BASC" survey | At 3 months after recruitment
  To evaluate the benefits of treatment at the neurocognitive level (Behavior Assesment)
Change in "BASC" survey | At 6 months after recruitment
  To evaluate the benefits of treatment at the neurocognitive level (Behavior Assesment)
Statistically significant changes in neuroimaging tests | At 3 months after recruitment
  Changes in structural imaging (white matter volume, gray matter volume and total intracranial volume, brain lobe volume and voxel-based morphometry), in diffusion (diffusion maps and structural connectivity) and in functional imaging (resting-state fMRI and task-based fMRI).
Statistically significant changes in neuroimaging tests | At 6 months after recruitment
  Changes in structural imaging (white matter volume, gray matter volume and total intracranial volume, brain lobe volume and voxel-based morphometry), in diffusion (diffusion maps and structural connectivity) and in functional imaging (resting-state fMRI and task-based fMRI).
Immune and inflammatory biomarkers | Baseline
  Study of lymphocyte populations by parametric flow cytometry (T lymphocytes, B lymphocytes, NK lymphocytes, NK T lymphocytes) and inflammatory cytokines by LUMINEX (IL-2, IL-4, IL-6, TNF alpha, IFN gamma, IL-10, IL-17a, IL-1R antagonist)
Statistically significant changes in immune and inflammatory biomarkers | At 3 months after recruitment
  Study of lymphocyte populations by parametric flow cytometry (T lymphocytes, B lymphocytes, NK lymphocytes, NK T lymphocytes) and inflammatory cytokines by LUMINEX (IL-2, IL-4, IL-6, TNF alpha, IFN gamma, IL-10, IL-17a, IL-1R antagonist)
Statistically significant changes in immune and inflammatory biomarkers | At 6 months after recruitment
  Study of lymphocyte populations by parametric flow cytometry (T lymphocytes, B lymphocytes, NK lymphocytes, NK T lymphocytes) and inflammatory cytokines by LUMINEX (IL-2, IL-4, IL-6, TNF alpha, IFN gamma, IL-10, IL-17a, IL-1R antagonist)

SECONDARY OUTCOMES:
Prevalence | Baseline
  To define the prevalence of neurocognitive deficit in cancer survivors in our population.
Perception of the family measured by satisfaction survey | Through study completion, 6 months
  To analyze the psychological and emotional perception of family members after a controlled intervention using video games.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Pérez-Martínez, PhD, Principal Investigator — Hospital la Paz
Locations (1):
- Hospital La Paz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol
Time Frame: Starting right after publication, for at least 1 year
Access Criteria: Sharing by personal contact

REFERENCES:
- [Background] Alonso Puig M, Alonso-Prieto M, Miro J, Torres-Luna R, Plaza Lopez de Sabando D, Reinoso-Barbero F. The Association Between Pain Relief Using Video Games and an Increase in Vagal Tone in Children With Cancer: Analytic Observational Study With a Quasi-Experimental Pre/Posttest Methodology. J Med Internet Res. 2020 Mar 30;22(3):e16013. doi: 10.2196/16013. PMID 32224482
- [Background] Argyriou AA, Assimakopoulos K, Iconomou G, Giannakopoulou F, Kalofonos HP. Either called "chemobrain" or "chemofog," the long-term chemotherapy-induced cognitive decline in cancer survivors is real. J Pain Symptom Manage. 2011 Jan;41(1):126-39. doi: 10.1016/j.jpainsymman.2010.04.021. Epub 2010 Sep 15. PMID 20832978
- [Background] Semendric I, Pollock D, Haller OJ, George RP, Collins-Praino LE, Whittaker AL. Impact of "chemobrain" in childhood cancer survivors on social, academic, and daily living skills: a qualitative systematic review protocol. JBI Evid Synth. 2022 Jan 1;20(1):222-228. doi: 10.11124/JBIES-21-00115. PMID 34341312
- [Background] Dovis S, Van der Oord S, Wiers RW, Prins PJ. Improving executive functioning in children with ADHD: training multiple executive functions within the context of a computer game. a randomized double-blind placebo controlled trial. PLoS One. 2015 Apr 6;10(4):e0121651. doi: 10.1371/journal.pone.0121651. eCollection 2015. PMID 25844638
- [Background] Gerbie MV. Management of the adolescent girl exposed in utero to DES. Pediatr Ann. 1981 Dec;10(12):23-6. PMID 7335401
- [Background] Conklin HM, Ogg RJ, Ashford JM, Scoggins MA, Zou P, Clark KN, Martin-Elbahesh K, Hardy KK, Merchant TE, Jeha S, Huang L, Zhang H. Computerized Cognitive Training for Amelioration of Cognitive Late Effects Among Childhood Cancer Survivors: A Randomized Controlled Trial. J Clin Oncol. 2015 Nov 20;33(33):3894-902. doi: 10.1200/JCO.2015.61.6672. Epub 2015 Oct 12. PMID 26460306
- [Background] Conklin HM, Ashford JM, Clark KN, Martin-Elbahesh K, Hardy KK, Merchant TE, Ogg RJ, Jeha S, Huang L, Zhang H. Long-Term Efficacy of Computerized Cognitive Training Among Survivors of Childhood Cancer: A Single-Blind Randomized Controlled Trial. J Pediatr Psychol. 2017 Mar 1;42(2):220-231. doi: 10.1093/jpepsy/jsw057. PMID 27342301
- [Background] Benzing V, Eggenberger N, Spitzhuttl J, Siegwart V, Pastore-Wapp M, Kiefer C, Slavova N, Grotzer M, Heinks T, Schmidt M, Conzelmann A, Steinlin M, Everts R, Leibundgut K. The Brainfit study: efficacy of cognitive training and exergaming in pediatric cancer survivors - a randomized controlled trial. BMC Cancer. 2018 Jan 3;18(1):18. doi: 10.1186/s12885-017-3933-x. PMID 29298678
- [Background] da Silva Alves R, Abdalla DR, Iunes DH, Mariano KOP, Borges JBC, Murta EFC, Michelin MA, Carvalho LC. Influence of an Exergaming Training Program on Reducing the Expression of IL-10 and TGF-beta in Cancer Patients. Games Health J. 2020 Dec;9(6):446-452. doi: 10.1089/g4h.2020.0022. Epub 2020 Jun 4. PMID 32498637
- [Background] Spitzhuttl JS, Kronbichler M, Kronbichler L, Benzing V, Siegwart V, Pastore-Wapp M, Kiefer C, Slavova N, Grotzer M, Roebers CM, Steinlin M, Leibundgut K, Everts R. Impact of non-CNS childhood cancer on resting-state connectivity and its association with cognition. Brain Behav. 2021 Jan;11(1):e01931. doi: 10.1002/brb3.1931. Epub 2020 Nov 18. PMID 33205895
- [Background] Lee H, Voss MW, Prakash RS, Boot WR, Vo LT, Basak C, Vanpatter M, Gratton G, Fabiani M, Kramer AF. Videogame training strategy-induced change in brain function during a complex visuomotor task. Behav Brain Res. 2012 Jul 1;232(2):348-57. doi: 10.1016/j.bbr.2012.03.043. Epub 2012 Apr 6. PMID 22504276
- [Background] Richlan F, Schubert J, Mayer R, Hutzler F, Kronbichler M. Action video gaming and the brain: fMRI effects without behavioral effects in visual and verbal cognitive tasks. Brain Behav. 2017 Dec 16;8(1):e00877. doi: 10.1002/brb3.877. eCollection 2018 Jan. PMID 29568680
- [Derived] Gonzalez-Perez C, Fernandez-Jimenez E, Moran E, Melero H, Malpica N, Alvarez-Linera J, Alonso Puig M, Plaza D, Perez-Martinez A. Study protocol for a randomized controlled clinical trial of a multifaceted cognitive training program using video games in childhood cancer survivors. PLoS One. 2025 Sep 2;20(9):e0314118. doi: 10.1371/journal.pone.0314118. eCollection 2025. PMID 40892751